CLINICAL TRIAL: NCT03282903
Title: The PRognostic Effect of Environmental Factors in Crohn's and Colitis
Acronym: PREdiCCt
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: University of Aberdeen (Other); Wellcome Sanger Institute (Other); NHS Lothian (Other Government); Chief Scientist Office of the Scottish Government (Other Government); Crohn's and Colitis in Childhood (Unknown); Cure Crohn's and Colitis (Unknown); Edinburgh and Lothain Health Fund (Lothian Health Board) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 16/WM/0152; IRAS183889 (Other: IRAS)
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample (for microbiome analysis) Saliva sample (for genomic analysis) Blood sample (for biochemical, haematological and genomic analysis)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's disease patients: 1550 Crohn's disease patients who are symptomatically controlled.
- Ulcerative Colitis patients: 1550 Ulcerative Colitis patients who are symptomatically controlled.

SUMMARY:
The PREdiCCt Study:

This is a major study that is now being launched. This is the first study of its kind and is specifically directed toward understanding how environmental factors and the gut microorganisms influence IBD flare and recovery. For the PREdiCCt study, the investigators hope to recruit 3100 people in remission from Crohn's disease or ulcerative colitis (illness under control) from 28 inflammatory bowel disease clinics across the UK.

The investigators hope to conduct the study in the following stages;-

1. Patients with Crohn's disease, ulcerative colitis or inflammatory bowel disease unclassified (IBDU) in clinical remission (under control) will be approached in gastroenterology clinics across the country and invited to take part in the PREdiCCt study. Alternatively they will express their interest in the study after seeing PREdiCCt promotional leaflets/posters/videos/social media.
2. Participants will attend a clinic visit for routine tests and also to complete several questionnaires with a research nurse.
3. At home over the next week participants will complete detailed questionnaires assessing their environment and diet. Participants will also collect a stool and saliva sample and send this to our laboratories (the investigators have developed easy ways of doing this reliably by post). The stool sample is to analyse the microorganisms in the participant's gut and the saliva is used to analyse their DNA. In addition to this the participants are asked to complete a 4-day weighed food diary. The food diary is sent to the University of Aberdeen for analysis.
4. Investigators will then follow patients' progress over 24 months. They will be asked to complete a short questionnaire every month with a longer questionnaire after 12 months and culminating in a final questionnaire 24 months after their initial clinic visit.
5. If a participant experiences a flare, investigators will collect an additional stool sample; but most importantly investigators will look to see how the environmental and microorganism factors recorded at the beginning differ for those that flare up versus those that don't.

What investigators hope to achieve;-

1. Finding out the environmental and dietary factors for patients to avoid because they trigger flare.
2. Finding out behaviours for patients to adopt because they bring about remission.
3. Finding out what the microorganisms that predict flare look like.
4. Gaining information which helps future studies aimed at finding better diets for IBD sufferers.
5. Developing ways of gathering information online from IBD patients about their well-being that doctors can routinely use.

The investigators have assembled expert doctors, epidemiologists, microbiologists, nutrition scientists, and bioinformaticians. These experts will use the systems the investigators have put in place to make sure PREdiCCt succeeds. It will yield a lot of new information to help sufferers right away; but the information will also help to kick start many important future studies that will bring us ever closer to a cure for Crohn's disease and ulcerative colitis.

DETAILED DESCRIPTION:
Background

Inflammatory bowel disease (IBD) is a common cause of chronic ill-health among young people in the UK (prevalence estimated at 1 in 200 for adults and 1 in 2000 for children, with a peak incidence in the second and third decades of life)1-2. The major forms of IBD, namely Crohn's disease (CD) and ulcerative colitis (UC), all too often confer a lifetime of unpleasant, intrusive and potentially dangerous burden of intestinal inflammation on individuals. Typical symptoms include abdominal pain, diarrhoea, weight loss, and lethargy. These adversely affect schooling, work attainment, psycho-social well-being and sexual health 3-4. IBD costs the NHS £720 million per year, based on an average per patient cost of £3,000; of which half of the costs are directly attributable to relapsing patients 5. Healthcare expenditure focus in IBD is shifting from hospitalisation and surgery to medical therapy 6. However, existing treatment modalities remain limited by lack of efficacy, unacceptable toxicity and poor patient acceptability. Major surgical intervention is frequently required (>50% in CD; ~20% in UC), with a high risk of disease recurrence, and there is an increased risk of cancer (in CD), with the highest incidence of colon cancer observed in those patients with poorly controlled disease 7. Nevertheless, there is a wide spectrum of disease severity. Around one third of patients will follow a relatively quiescent disease course 8. Understanding who gets severe, progressive disease and why, is an urgent research priority. Accurate prediction of these patients will enable precise, tailored intervention early in the disease course. This should reduce the substantial morbidity and costs associated with IBD.

Genetics, Environment and the Microbiota and Disease Natural History.

Genetic factors play a modest role in defining disease location and extent but not disease behaviour 9-12. There is very limited evidence about the gut microbiota in disease progression, although emerging data support a potential role in treatment response. We cannot alter our genes and, despite intense interest in modifying the gut microbiota (e.g. faecal transplantation) there is only limited clinically data to support this 13-14. However, it is within our control to change what we eat and to therefore potentially modify our gut microbiota to a more favourable phenotype. Patients suspect this should be part of the answer: one of the commonest questions in the clinic is, "What should I eat?" Established clinical strategies include the use of exclusive enteral nutrition (EEN) to induce remission in CD, and a low fibre diet to alleviate obstructive symptoms in stricturing disease 15. However, beyond this there is presently very limited data to support any on-going specific dietary strategy for the vast majority of patients with IBD 16. Multiple lines of emerging evidence in animal models suggest that diets high in natural plant fibres favour an anti-inflammatory gut milieu, via alterations in the gut microbiota, measurable by short-chain fatty acid (SCFA) concentrations in stool 17. Dietary fibre may protect against the development of IBD, through several mechanisms, through its conversion to acetate, butyrate and propionate (the major SCFAs). Firstly, butyrate is the main energy source for colonocytes and is associated with the maintenance of the intestinal epithelium 18. Secondly, SCFAs have immunomodulatory roles including inhibition of the transcription factor NF-KB and are the only known ligands of G-protein-coupled receptor, GPR43, which limits the inflammatory response 19-20. Interestingly, the fermentation of fibre is dependent on gut microbiota, such as Bacteroidetes species, which are deficient in patients with IBD 21. The individual source of fibre may also be important. In the US Nurses' Health Study of 170,776 women with 3,317,425 person-years of follow-up over 26 years there were 269 incident cases of Crohn's disease diagnosed and 338 cases of ulcerative colitis 22. For the latter illness, there were no associations with either total dietary fibre intake or fibre from any specific food groups. However, for Crohn's disease the highest quintile of energy-adjusted cumulative average dietary fibre intake, namely 24.3 g/day, was associated with a 41% reduction in risk compared with the lowest quintile (hazard ratio (HR) =0.59, 95% confidence interval (CI=)=0.39-0.90). This reduction was associated with the fibre content from fruits (highest vs. lowest quintile HR=0.57, 95% CI=0.38-0.85) with no associations detected between fibre from vegetables, cereals or legumes.

These are important issues; the lack of data means patients may resort to untested and potentially harmful 'fad' diets 16. More pressingly, this is potentially a novel therapeutic approach to both induce and maintain prolonged remission. Interventional studies in cases and controls will be necessary, but first further data are required from observational epidemiological studies to inform which 'interventions' are indicated and/or justified.

Rationale for the Study

It is presently very hard to predict which IBD patients in remission will flare and when. Scant data are available to advise patients on any substantial lifestyle measure they can adopt to help prevent or retard future disease from flaring. Potential areas of direct relevance to patients are aspects of habitual diet, regular exercise, sleep and stress, including that from major life events. It is hypothesised that there are multiple factors in habitual diet that are associated with increased risk of disease flare, including reduced levels of dietary fibre, high levels of n-6 PUFAs, low levels of n-3 PUFAs and dietary emulsifiers. High levels of regular physical activity are also hypothesised to reduce the rates of disease flare. These dietary aspects and facets in concert with other lifestyle factors may contribute in part to the intestinal dysbiosis associated with flare, where the investigators anticipate seeing a reduction in microbial diversity.

The major aim of this study is to identify the environmental and gut microbiota factors that predispose to disease flare and influence disease outcomes in IBD. Further, the investigators aim to build intelligent predictive models of disease behaviour and prognosis combining phenotypic, environmental and biological data inputs of direct clinical utility.

ELIGIBILITY:
Inclusion Criteria:

- Confirmed Crohn's disease or ulcerative colitis or IBDU (Lennard-Jones/Porto criteria).

Clinical remission (see definition Section 3.2 of protocol) >6 months since diagnosis with Crohn's disease, ulcerative colitis or IBDU >2 months since any change in therapy for Crohn's disease, ulcerative colitis or IBDU Aged six years or over at study entry Written informed consent obtained from patient or parent / guardian

Exclusion Criteria:

- Patient unwilling to take part in all aspects of the study Unable to obtain written informed consent Systemic corticosteroids (oral or intravenous) within the last two months Thiopurines / methotrexate / biologic therapy started in the preceding two months

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IBD patients with a confirmed diagnosis of Crohn's Disease, Ulcerative Colitis or IBD unspecified, who are in clinical remission, >6 since diagnosis, >2 months since any change in therapy for Crohn's disease, ulcerative colitis or IBDU, aged 6 or over at study entry and who informed consent can be obtained from (or parent/guardian).
Sampling Method: Non-Probability Sample
Enrollment: 2629 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Clinical flare | Up to 2 years
  Patients will be asked to answer a monthly follow up, providing details of their IBD over the last month. A clinical flare will be determined by a patient answering "no" to the following question in the monthly follow up:
  "Do you think your disease has been well controlled in the past 1 month?"

SECONDARY OUTCOMES:
Hard clinical flare | Up to 2 years
  Clinical flare (primary outcome) plus commencement of any new medication; altered dosing of existing medication for the treatment of IBD flare, with an increase in CRP (>5mg/L) and / or faecal calprotectin (>200mcg/g).

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Lees, Principal Investigator — University of Edinburgh
Locations (41):
- United Kingdom (41):
  - Aberdeen Royal Infirmary, Aberdeen
  - Bronglais General Hospital, Aberystwyth
  - NHS Lanarkshire, Airdrie
  - Ulster Hospital, Belfast
  - Bristol Royal Infirmary, Bristol
  - West Suffolk NHS Foundation Trust, Bury St Edmunds
  - Cambridge Addenbrooke's Hospital, Cambridge
  - Glangwili General Hospital, Carmarthen
  - University Hospital Coventry & Warwickshire, Coventry
  - Darlington Memorial Hospital, Darlington
  - Ninewells Hospital, Dundee
  - Eastbourne General Hospital, Eastbourne
  - Western General Hospital, Edinburgh
  - Royal Hospital for Sick Children,Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Queen Elizabeth Hospital, Gateshead
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Royal Hospital for Children, Glasgow, Glasgow
  - Withybush General Hospital, Haverfordwest
  - Raigmore Hospital, Inverness
  - Kettering General Hospital NHS Foundation Trust, Kettering
  - Queen Elizabeth King's Lynn, Kings Lynn
  - Kingston Hospital, Kingston upon Thames
  - NHS Fife, Kirkcaldy
  - NHS Forth Valley, Larbert
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool
  - St John's Hospital, Livingston
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Royal Free Hospital, London
  - Royal London Hospital (Barts Health), London
  - Newcastle Royal Victoria Hospital, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Royal Berkshire Hospital, Reading
  - Salford Royal Hospital, Salford
  - Sandwell and West Birmingham Hospitals NHS Trust, Sandwell
  - Buckinghamshire Healthcare NHS Trust, Stoke Mandeville
  - Musgrove Park Hospital, Taunton
  - Pinderfield General Hospital, Wakefield
  - Warrington and Halton NHS FT, Warrington
  - Royal Hampshire Hospital, Winchester

IPD SHARING:
Plan to Share IPD: No
Anonymised data will be shared with collaborators to allow analysis.
  Only aggregate level data will be published.

REFERENCES:
- [Derived] Constantine-Cooke N, Gros B, Plevris N, Williams LJ, Jones GR, Kyle J, Kennedy NA, Velasco-Pardo V, Rudge A, Alexander D, Anderson CA, Brusco de Freitas M, Derr LM, Derikx LA, Gilchrist S, Henderson P, Horgan GW, Irving P, Lamb CA, Jostins-Dean L, Lindsay JO, MacDonald J, Mowat C, Murray C, Parkes M, Siakavellas SI, Vallejos CA, Gaya DR, Rhodes JM, Johnstone AM, Weir CJ, Lees CW; PREdiCCt study group. Associations between demographic, clinical and dietary factors and flares in inflammatory bowel disease: the PRognostic effect of Environmental factors in Crohn's and Colitis (PREdiCCt) prospective cohort study. Gut. 2026 Jan 19:gutjnl-2025-337846. doi: 10.1136/gutjnl-2025-337846. Online ahead of print. PMID 41554630